CLINICAL TRIAL: NCT01583023
Title: Assessing the Efficacy of Left Repetitive Transcranial Magnetic Stimulation (rTMS) as an Adjunctive Treatment to Mood Stabilizers for the Treatment of Bipolar Depression
Brief Title: Using Repetitive Transcranial Magnetic Stimulation (rTMS) for the Treatment of Bipolar Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Pablo Cervantes, Director of the Mood Disorders Clinic, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RTMS-BD-1
Record Dates: First submitted 2012-04-19; First posted 2012-04-23 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; repetitive transcranial magnetic stimulation (rtms); bupropion; lithium a/o Epival
MeSH Terms: conditions — Bipolar Disorder | interventions — Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wellbutrin + Lithium a/o Epival + Sham rTMS (Experimental)
  Interventions: Drug: Bupropion; Device: Sham repetitive transcranial magnetic stimulation
- Placebo + Lithium a/o Epival + Active rTMS (Experimental)
  Interventions: Device: Active Repetitive Transcranial Magnetic Stimulation; Other: Placebo
- Wellbutrin + Lithium a/o Epival + Active rTMS (Experimental)
  Interventions: Drug: Bupropion; Device: Active Repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Drug: Bupropion — 150mg daily for first week, 300mg daily thereafter for a total of 8 weeks
  Other Names: Wellbutrin
  Arms: Wellbutrin + Lithium a/o Epival + Active rTMS; Wellbutrin + Lithium a/o Epival + Sham rTMS
Device: Active Repetitive Transcranial Magnetic Stimulation — Daily left DLPFC, at 110% motor threshold, with a frequency of 10 Hz. Stimulation will be applied in 5-second trains with a 10-second inter-train interval, for 30 trains per session. This treatment will be provided for the first 4 weeks of the study.
  Arms: Placebo + Lithium a/o Epival + Active rTMS; Wellbutrin + Lithium a/o Epival + Active rTMS
Other: Placebo — 150mg daily first week, 300mg daily thereafter for a total of 8 weeks.
  Arms: Placebo + Lithium a/o Epival + Active rTMS
Device: Sham repetitive transcranial magnetic stimulation — Sham rTMS will also begin their treatment 5 times a week for 4 weeks in junction with pharmacotherapy (Wellbutrin). Sham rTMS will be delivered at a frequency of 10 Hz and stimulation will be applied in 5-second trains with a 20-second inter-train interval, for 30 trains per session.
  Arms: Wellbutrin + Lithium a/o Epival + Sham rTMS

SUMMARY:
The purpose of this study is to evaluate whether repetitive transcranial magnetic stimulation (rTMS) treatment is an effective adjunct treatment to mood stabilizers and Bupropion.

ELIGIBILITY:
Inclusion Criteria:

BD Type I or II subjects diagnosed according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) in depressed phase.

Age 18 to 70. Rating on the Montgomery-Asberg Depression Rating Scale (MADRS) score > 20. Rating on the Beck Depression Inventory (BDI-II) > 20. Rating on the Young Mania Rating Scale (YMRS) < 8. Non-treated new depressive episode, at least 2 weeks in duration. If recently started on an antidepressant other than Wellbutrin, subject must spend at least 4 weeks at a therapeutic dose before entering the study.

Lithium and epival (Sodium Valproate) in monotherapy or in combination. Novel antipsychotics can be combined with mood stabilizers for at least 4 weeks at a steady dosage prior to the study.

Exclusion Criteria:

History of any DSM-IV Axis I diagnosis other than BD Type I or II Presence of any psychotic symptoms, characterized by a score of 3 or more on item 10 of the MADRS, a score of 6 on item 9 of the MADRS, or a score of 6 or more on item 8 of the YMRS Comorbid active dependence or substance abuse (except nicotine) Prior electroconvulsive therapy failure Pacemaker, automatic implantable defibrillator or implantable pump Aneurysm Clip Heart/Vascular Clip Prosthetic Valve Metal Prosthesis Pregnancy (must do a blood β-HCG test to exclude) Metal or metal fragments in the head Personal or Family history of seizure disorder Increased Intracranial pressure History of stroke, meningitis/encephalitis, moderate to severe traumatic brain injury, neurosurgical procedure Pharmacotherapy using any substances not mentioned in the inclusion criteria, except benzodiazepines at an equivalent dose of less than or equal to 1mg/day of lorazepam.

Failure of previous Wellbutrin treatment. Mood disorder secondary to a medical condition. Subject currently enrolled in any detoxification program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale (MADRS) from baseline at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
Change in Beck Depression Inventory (BDI-II) from baseline at 8 weeks | 8 weeks
Change in Young Mania Rating Scale (YMRS) from baseline at 8 weeks | 8 weeks
Alcohol use disorder identification test (AUDIT Assessment) | At intake
Drug abuse screen test (DAST Assessment) | At intake
Clinical Global Impression (CGI) & Analog scale | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Cervanes, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Theodore Kolivakis, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Nancy CP Low, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Gabriella Gobbi, M.D, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Allan Memorial Institute, Montreal, Quebec, Canada